CLINICAL TRIAL: NCT02044224
Title: Effects of Dexmedetomidine on Anaesthesia During IRE Procedures for Solid Tumours
Brief Title: Effects of Dexmedetomidine During IRE Procedures for Solid Tumours
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Egidijus Semenas, Consultant in anaesthesia and intensive care, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRE-01; 2013/413 (Other: Uppsala Regional Ethics Committe)
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Cancer of Liver; Cancer of Pancreas
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomidine (Experimental): Dexmedetomidine infusion during anaesthesia for IRE procedure
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.4 µg/kg/hr infusion (from the start of anaesthesia until the end of anaesthesia).
  Anaesthesia induction: propofol 2 mg/kg, rocuronium 0.6 mg/kg iv, and fentanyl 2-3 mikrogram/kg.
  Anaesthesia maintenance: sevoflurane and oxygen 50%, rocuronium 0.1-0.2 mg/kg iv, fentanyl 1 mikrogram/kg as required

SUMMARY:
The purpose of the study is to evaluate effects of dexmedetomidine on anaesthesia during IRE procedures for solid tumours

DETAILED DESCRIPTION:
Pulsed electric current can be used to produce irreversible electroporation (IRE) of cell membranes with resulting cell death. This process has been shown to ablate tumors in animal and human studies. A pulsating direct current of 20 to 50 A and 500 to 3000 V is delivered into metastatic or primary tumors in the liver, kidney, or lung via needle electrodes inserted under computed tomography (CT) or ultrasound guidance. Patients usually require general anesthesia with muscle relaxant. Currently, circa 30 procedures have been done at our institution with good or excellent results. However, several patients have had severe pain postoperatively.

Dexmedetomidine is an α2-adrenoreceptor agonist with sedative, analgesic and anxiolytic effects, and it has more selective α2-adrenergic effect than clonidine. We will evaluate perioperative dexmedetomidine 0.4 µg/kg/hr infusion effects on hemodynamics, anesthetic consumption, and recovery profiles during anesthesia for IRE of solid organs tumours.

ELIGIBILITY:
Inclusion Criteria:

1. liver or/and pancreas cancer for which IRE procedure is planned
2. signed informed consent form

Exclusion Criteria:

1. patient refusal
2. pregnancy
3. known allergy to dexmedetomidine or other anaesthesia drugs
4. atrioventricular block grade II or III or other significant cardiac conduction disturbance
5. stroke
6. low blood pressure not responding to treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction With Anaesthesia Technique | At the discharge from post-anaesthesia care room (up to 4 hours after the procedure)
  Rating of how satisfied the patient was with their sedation on a scale of 1-5 with 1 being very dissatisfied and 5 being extreme

SECONDARY OUTCOMES:
Evaluation of anaesthetic consumption | During anaesthesia
Vital signs: blood pressure, oxygen saturation, heart rate, breathing rate | During procedure and up to 4 hours stay at the post-anesthesia care unit
Postoperative analgesic requirements | During the first 24 hours after procedure
Maximal pain intensity | During stay at the post-anesthesia care unit (up to 4 hr) and during the first 24 hours after procedure
  The 11-point Numerical Rating Scale (NRS) to assess periprocedural pain. Scale of 0-10, with 0:no pain and 10: pain as bad as it could be
Description of patient characteristics | During one week before preoperative visit at anaesthesia clinic
  Primary disease, concomitant diseases, medications, allergies

CONTACTS AND LOCATIONS:
Overall Officials: Egidijus Semenas, MD, PhD, Principal Investigator — Uppsala University Hospital, Uppsala, Sweden; Mats Eriksson, MD, PhD, Principal Investigator — Uppsala University Hospital, Uppsala, Sweden
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] Jones CR. Perioperative uses of dexmedetomidine. Int Anesthesiol Clin. 2013 Spring;51(2):81-96. doi: 10.1097/AIA.0b013e31828d58c7. No abstract available. PMID 23532129
- [Background] Yazbek-Karam VG, Aouad MM. Perioperative uses of dexmedetomidine. Middle East J Anaesthesiol. 2006 Oct;18(6):1043-58. No abstract available. PMID 17263262
- [Background] Barletta JF, Miedema SL, Wiseman D, Heiser JC, McAllen KJ. Impact of dexmedetomidine on analgesic requirements in patients after cardiac surgery in a fast-track recovery room setting. Pharmacotherapy. 2009 Dec;29(12):1427-32. doi: 10.1592/phco.29.12.1427. PMID 19947802
- [Background] Cheung W, Kavnoudias H, Roberts S, Szkandera B, Kemp W, Thomson KR. Irreversible electroporation for unresectable hepatocellular carcinoma: initial experience and review of safety and outcomes. Technol Cancer Res Treat. 2013 Jun;12(3):233-41. doi: 10.7785/tcrt.2012.500317. Epub 2013 Jan 25. PMID 23369152
- [Background] Ball C, Thomson KR, Kavnoudias H. Irreversible electroporation: a new challenge in "out of operating theater" anesthesia. Anesth Analg. 2010 May 1;110(5):1305-9. doi: 10.1213/ANE.0b013e3181d27b30. Epub 2010 Feb 8. PMID 20142349